CLINICAL TRIAL: NCT04146649
Title: Effect of Therapeutic Joint Arthrocentesis on Pain and Quadriceps Function in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Jason Jennings, Primary Investigator, Colorado Joint Replacement
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1415301
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Effusion Joint
MeSH Terms: conditions — Hydrarthrosis | interventions — Arthrocentesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Osteoarthritis (Experimental): Patients with native knees and effusions will participate in this arm.
  Interventions: Procedure: Arthrocentesis
- Primary TKA (Experimental): Patients with total knee replacements will participate in this arm.
  Interventions: Procedure: Arthrocentesis

INTERVENTIONS:
Procedure: Arthrocentesis — Patients will receive a joint arthrocentesis to remove fluid from the joint.

SUMMARY:
This will be prospective study of patients with knee effusion associated with degenerative osteoarthritis or symptomatic primary total knee arthroplasty that undergo therapeutic joint arthrocentesis. The diagnosis of knee osteoarthritis will be based on knee radiographs (including AP, Rosenburg view, lateral and Merchant views) read and interpreted by one of our clinical providers (PA, Fellow or Surgeon). Patients with at least Grade II Kellgren and Lawrence changes or higher will be included in the osteoarthritis group. Patients in the arthroplasty group must have had a primary total knee arthroplasty without infection (as determined by knee aspirate) to be included. Patients will be clinically evaluated at the time of their visit for presence of a knee effusion using a stroke test and graded on a 5-point scale (zero, trace, 1+, 2+, or 3+) which has shown good interrater reliability. Patients with a mild to severe effusion (1+ to 3+) will considered for the study. Patients having significant pain associated with their effusion will be offered a therapeutic arthrocentesis as part of their treatment plan discussion. This is a pre-post test design in which outcome measures will be collected immediately pre-arthrocentesis and immediately post arthrocentesis. Additionally, there will be an optional 7-10 follow up visit where outcomes measures will be collected again, should the participant choose to return to this visit.

DETAILED DESCRIPTION:
Pain and Self-Reported Function

Knee pain will be assessed with an 11-point numeric pain rating scale (NPRS) where 0 represents 'no pain' and 10 represents 'worst imaginable pain'. Self-reported physical function will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for each knee separately. The WOMAC assesses the impact of knee osteoarthritis on multiple domains-pain, stiffness, and disability. A composite score (0-100 scale) will be used for analysis.

Range of Motion

Knee range of motion (ROM) is a direct measure of joint mobility following TKA. Knee ROM will be measured in the supine position both actively and passively using a long-arm goniometer. Goniometry has been shown to be a reliable measure of knee ROM after TKA.

Quadriceps Strength and Activation Testing

Maximum voluntary isometric quadriceps strength and quadriceps activation will be assessed before surgery and at week 3 using an electromechanical dynamometer (Humac Norm, CSMI) and a doublet interpolation test. Patients will be seated on the electromechanical dynamometer with their hips flexed to approximately 85° and their knees flexed to 60°. Two 3" by 5" self-adhesive neuromuscular stimulation electrodes will be placed over the motor points of the rectus femoris and the vastus medialis. A Grass S48 stimulator with a Grass Model SIU8T stimulus isolation unit will be used to deliver 600 µs doublet pulses. A Biopac MP150WSW system will be used for data acquisition during testing with sampling frequency of 300 Hz.

Following two warm-up contractions, a practice maximal voluntary isometric contraction (MVIC) will be performed against the dynamometer's force transducer. Visual torque targets will be set on the feedback monitor at slightly higher torques than produced during the practice MVIC trial. Trials will be repeated until maximal torque is within 5% of the previous attempt. Torque from quadriceps MVIC will be normalized to body weight for between-subject comparisons.

Voluntary activation of the quadriceps muscle will be assessed using the doublet interpolation technique, where a supramaximal stimulus will be applied by a Grass S48 stimulator during an MVIC and immediately afterwards while the quadriceps muscle is at

rest. Normalization of the force from the superimposed doublet to the resting doublet allows for comparisons of quadriceps activation across individuals and lower extremities.

Timed-Up-and-Go

The timed-up-and-go (TUG) test is a responsive, valid, and reliable functional measure of basic mobility and dynamic balance. The examiner measures the time, in seconds, required by the patient to a) rise from an arm chair; b) walk 3 meters; c) turn and walk back to the arm chair; and d) return to the seated position.

30-second Sit-to-Stand Test

The 30-second Sit-to-Stand test (30STS) is a responsive, valid, and reliable functional measure of lower extremity strength after TKA. This test counts the number of times a patient can rise to a full standing position in 30 seconds. The test starting position is sitting on an armless chair with seat plate 17 inches from the floor. Patients rise from this position with hands placed on opposite shoulders. If the patient must use his/her arms to stand, the test is stopped. If the patient is over halfway to a standing position when 30 seconds have lapsed, this counts as a stand.

Bioimpedance Spectroscopy

Bioimpedance spectroscopy (BIS) is a reliable, responsive measure of swelling that has been validated in observational studies of individuals after TKA. The RJL Systems Quantum® (Clinton Township, MI) bioelectrical impedance device delivers a 2.5 µA alternating current at a frequency of 50 kHz. The tissue impedance to this current is displayed in Ohms (Ω) and is recorded at a precision of 1 Ω. The level of impedance met by the current reflects the composition of the tissue, but will also fluctuate with the presence of swelling in the lower extremity. Lower levels of impedance represent the increased fluid content present with greater levels of swelling. Measuring the impedance of both the involved and uninvolved limb allows for calculation of a ratio (W-involved limb: W-uninvolved limb). To measure impedance, a four-wire measurement method will be used. The most proximal electrode pair will be placed 10 and 20 centimeters above the superior patellar pole. The most distal electrode pair will be placed at a point bisecting the medial and lateral malleolus, and also 10 cm distal to that point along the second ray of the foot. New electrodes will be used for each testing session, and skin will be cleaned with an alcohol swab prior to electrode placement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older with mild (1+) to severe (3+) knee effusion associated with underlying osteoarthritis (Kellgren and Lawrence grade II or higher) that undergo therapeutic aspiration
2. Patients with symptomatic primary total knee arthroplasty without infection (as verified by prior aspiration) with moderate to severe effusion electing for therapeutic arthrocentesis. Must be minimum of 3 months from index surgery to be included.

Exclusion Criteria:

1. Patients with effusion related to trauma or another underlying condition (ie. fracture, ligamentous injury, hemarthrosis)
2. Patients with known history of gout or with synovial fluid samples testing positive for urate of calcium pyrophosphate crystals
3. Patients with knee effusion associated with septic arthritis or periprosthetic knee infection as determined from knee arthrocentesis.
4. Patients with inflammatory arthritis (ie. JIA, RA, psoriatic arthritis, etc).
5. Patients with revision knee arthroplasty, unicompartmental arthroplasty or other repair/reconstruction surgery
6. Patients with underlying muscular disorder (ie. Stroke, cerebral palsy, multiple sclerosis, polymyalgia, fibromyalgia, muscular dystrophy, etc.)
7. Patients with symptomatic hip pain
8. Patients with active cancer in the area
9. Patients with pacemakers
10. Patients who are pregnant
11. Invasive or injectable therapy within the last 6 months in the involved knee, to include, but not limited to, arthrocentesis, corticosteroid, hyaluronic acid, platelet-rich plasma, prolotherapy, stem cell therapy, or genicular nerve block.
12. Blood clotting disorders, sickle cell disease or trait, or chronic anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps activation | Immediately pre aspiration (day 0), immediately post aspiration (day 0),optional 7-10 days post aspiration
  The change in quadriceps activation prior to and post arthrocentesis will be measured.

SECONDARY OUTCOMES:
Change in Pain | Immediately pre aspiration (day 0), immediately post aspiration (day 0), optional 7-10 days post aspiration
  Self reported pain scores
Function | Immediately pre aspiration (day 0), immediately post aspiration (day 0), optional 7-10 days post aspiration
  Self reported function will be collected
Range of Motion | Immediately pre aspiration (day 0), immediately post aspiration (day 0), optional 7-10 days post aspiration
  Range of motion will be measured
Quadriceps Strength | Immediately pre aspiration (day 0), immediately post aspiration (day 0), optional 7-10 days post aspiration
  This will be measured using the Humac Norm chair
Functional Performance | Immediately pre aspiration (day 0), immediately post aspiration (day 0), optional 7-10 days post aspiration
  This will be assessed with standardized functional tests (30 STS, TUG)
Volume of Knee Synovial Fluid Aspirated | Immediately post aspiration (day 0)
  We will look at the volume of fluid drawn off the knee
Bioelectrical Impedance | Immediately pre aspiration (day 0), immediately post aspiration (day 0), optional 7-10 days post aspiration
  This will be measured with The RJL Systems Quantum®

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jennings, MD, Principal Investigator — Colorado Joint Replacement
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Colorado Joint Replacement, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and most common causes of disability among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2009 May 1;58(16):421-6. PMID 19407734
- [Background] Neogi T. The epidemiology and impact of pain in osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1145-53. doi: 10.1016/j.joca.2013.03.018. PMID 23973124
- [Background] Dieppe PA, Lohmander LS. Pathogenesis and management of pain in osteoarthritis. Lancet. 2005 Mar 12-18;365(9463):965-73. doi: 10.1016/S0140-6736(05)71086-2. PMID 15766999
- [Background] Egloff C, Hugle T, Valderrabano V. Biomechanics and pathomechanisms of osteoarthritis. Swiss Med Wkly. 2012 Jul 19;142:w13583. doi: 10.4414/smw.2012.13583. eCollection 2012. PMID 22815119